CLINICAL TRIAL: NCT06171698
Title: Prospective Measurement of Impedance During Cardiac Catheterization to Build a Non-Invasive Cardiac Output Algorithm
Brief Title: Impedance During Cardiac Catheterization to Build a Non-Invasive Cardiac Output Algorithm
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed at site. Investigator no longer at location.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00281586
Record Dates: First submitted 2023-11-28; First posted 2023-12-15 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Research Prototype Monitor (Experimental)
  Interventions: Device: Research Prototype Monitor

INTERVENTIONS:
Device: Research Prototype Monitor — Continuous vital sign is collected via a research prototype monitor

SUMMARY:
Prospectively measure impedance during cardiac catheterization to build a cardiac output algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo cardiac catheterization with cardiac output measurement and Fick
* Planned to undergo general anesthesia for cardiac catheterization standard of care
* Parent/Guardian able to provide informed consent

Exclusion Criteria:

* Not planned for standard of care general anesthesia for cardiac catheterization

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Feasibility of a non-invasive monitoring device | From device placement to removal, up to 12 hours
  Feasibility of a non-invasive monitoring device that can accurately measure cardiac output in patients with congenital heart disease as determined by percent error compared to catheter-measured cardiac output.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Gottlieb Sen, MD, MPH, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Children's Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No